CLINICAL TRIAL: NCT05769504
Title: Studying Patient Experiences in Small Cell Lung Cancer Clinical Trials to Identify Influencing Factors
Brief Title: Examining Clinical Trial Participation for Small Cell Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 86382894
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical trial may make it more difficult for patients to take part or see it through.

The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future small cell lung cancer patients during clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Participant has a diagnosis of small cell lung cancer.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Pregnant or lactating woman
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Small cell lung cancer patients who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a small cell lung cancer clinical study. | 3 months
Number of small cell lung cancer patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Meerbeeck JP, Fennell DA, De Ruysscher DK. Small-cell lung cancer. Lancet. 2011 Nov 12;378(9804):1741-55. doi: 10.1016/S0140-6736(11)60165-7. Epub 2011 May 10. PMID 21565397
- [Background] Seto Z, Takata N, Murayama N, Tokui K, Okazawa S, Kambara K, Imanishi S, Miwa T, Hayashi R, Matsui S, Inomata M. Irinotecan monotherapy as third- or further-line treatment for patients with small cell lung cancer. Tumori. 2021 Dec;107(6):536-541. doi: 10.1177/0300891620974762. Epub 2020 Nov 25. PMID 34847814
- [Background] Xing H, Zhang J, Ge F, Yu X, Bian H, Zhang F, Fang J. [Analysis of the Efficacy of Irinotecan in the Second-line Treatment of Refractory and Relapsed Small Cell Lung Cancer]. Zhongguo Fei Ai Za Zhi. 2021 Mar 20;24(3):167-172. doi: 10.3779/j.issn.1009-3419.2021.103.04. Chinese. PMID 33819966

DOCUMENTS (1):
  • Informed Consent Form (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT05769504/ICF_000.pdf